CLINICAL TRIAL: NCT07321639
Title: Comparison of the Effectiveness of Ultrasound-Guided Recto-Intercostal Fascial Plane Block and Transversus Abdominis Plane Block in Postoperative Analgesia Management of Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Ultrasound-Guided Regional Blocks for Postoperative Analgesia After Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ayse Ince, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 7
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Laparoscopic Cholecystectomy; Acute Pain; Pain Management; Plane Blocks
Keywords: Laparoscopic cholecystectomy; Postoperative analgesia; Recto-intercostal fascial plane block; Transversus abdominis plane block; Regional anesthesia; Opioid consumption
MeSH Terms: conditions — Acute Pain; Agnosia | interventions — 1,3-bis(4-amidinophenoxy)-2-(4-amidinophenoxymethyl)ethylpropane

STUDY DESIGN:
Intervention Model Description: Ninety patients aged 18-65 years with American Society of Anesthesiologists (ASA) physical status I-II who are scheduled to undergo laparoscopic cholecystectomy will be included in the study. Patients will be randomly assigned to three groups before entering the operating room: the recto-intercostal fascial plane block group (Group RIFPB), the transversus abdominis plane block group (Group TAPB), and the control group, with 30 patients in each group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes assessor and participants will be blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recto-intercostal fascial plane block (Active Comparator): RIFP block will be performed, and standard postoperative pain management protocols will be applied.
  Interventions: Procedure: Recto-Intercostal Fascial Plane Block; Other: Post-operative Pain Management
- Transversus abdominis plane block (Active Comparator): TAP block will be performed, and standard postoperative pain management protocols will be applied.
  Interventions: Procedure: Transversus- Abdominis Plane Block; Other: Post-operative Pain Management
- Control group (Active Comparator): Standard postoperative pain management protocols will be applied. No plane block will be applied.
  Interventions: Other: Post-operative Pain Management

INTERVENTIONS:
Procedure: Recto-Intercostal Fascial Plane Block — The block will be performed under general anesthesia immediately before extubation, with the patient in the supine position under ultrasound guidance (Vivid Q). After aseptic preparation, a high-frequency linear probe (11-12 MHz) covered with a sterile sheath and an 80-mm block needle (Braun 360°) will be used. The probe will be positioned to identify the xiphoid process, rectus abdominis muscle, and sixth costal cartilage. Using an in-plane technique, the needle will be advanced in a caudal-to-cephalic direction. After confirmation of correct needle placement with 5 mL saline, 20 mL of 0.25% bupivacaine (Buvacaine, Polifarma ®) will be injected on each side (total volume 40 mL).
  Other Names: RIFPB
  Arms: Recto-intercostal fascial plane block
Procedure: Transversus- Abdominis Plane Block — The transversus abdominis plane block will be performed immediately after completion of surgery and before extubation, with the patient in the supine position under ultrasound guidance( Vivid Q). Following aseptic preparation, a high-frequency linear probe (11-12 MHz) and an 80-mm block needle (Braun 360°) will be used to identify the abdominal wall muscle layers at the anterior axillary line between the 12th rib and the iliac crest. Using an in-plane technique, the needle will be advanced into the plane between the internal oblique and transversus abdominis muscles. After confirmation of correct needle placement with 5 ml saline injection, 20 mL of 0.25% bupivacaine (Buvacaine, Polifarma ®) will be administered to each side (total volume 40 mL).
  Other Names: TAPB
  Arms: Transversus abdominis plane block
Other: Post-operative Pain Management — Thirty minutes before the end of surgery, all patients will receive the standard postoperative analgesia regimen consisting of intravenous ibuprofen 400 mg (Intrafen®) and intravenous tramadol 100 mg (Contramal®). Postoperative patient assessment will be performed by an anesthesiologist who is not involved in the intervention.If the patient's NRS score is ≥4 at any time point, intravenous meperidine (Aldolan®) at a dose of 0.5 mg/kg will be administered as rescue analgesia.

SUMMARY:
Ultrasound (US)-guided recto-intercostal fascial plane block (RIFPB) is a recently described abdominal wall block performed by injecting local anesthetic between the rectus abdominis muscle and the costal cartilage of the 7th rib. Due to the cranial attachment of the rectus muscle, this technique provides effective analgesia to the sternal, epigastric, and upper-mid abdominal regions, corresponding to the T6-T10/11 dermatomal levels. RIFPB may be used as an adjunct technique for thoracic procedures or as a standalone block for abdominal surgery.

Ultrasound-guided transversus abdominis plane block (TAPB) is performed by injecting local anesthetic into the fascial plane between the internal oblique and transversus abdominis muscles. TAPB provides sensory blockade of the anterolateral abdominal wall at the T6-L1 dermatomal levels and is widely used for postoperative analgesia following abdominal surgeries, including laparoscopic cholecystectomy.

This study aims to compare the effectiveness of US-guided RIFPB and TAPB on postoperative pain control after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is one of the most commonly performed abdominal surgical procedures. Postoperative pain after laparoscopic cholecystectomy is multifactorial and may result from trocar site incisions, visceral manipulation, peritoneal irritation, and diaphragmatic stimulation due to pneumoperitoneum. Various analgesic strategies, including systemic opioids, non-opioid analgesics, local anesthetic infiltration, and regional anesthesia techniques, are used to manage postoperative pain in these patients.

Ultrasound (US)-guided recto-intercostal fascial plane block (RIFPB) is a recently described regional anesthesia technique that provides analgesia to the sternal, epigastric, and upper-mid abdominal regions by targeting the fascial plane between the rectus abdominis muscle and the costal cartilage. RIFPB provides sensory blockade at the T6-T10/11 dermatomal levels and has been reported to be effective for postoperative analgesia in thoracic and upper abdominal procedures. Due to its anatomical spread and mechanism of action, RIFPB may offer effective analgesia following laparoscopic cholecystectomy.

Ultrasound-guided transversus abdominis plane block (TAPB) is a well-established regional anesthesia technique performed by injecting local anesthetic between the internal oblique and transversus abdominis muscles. TAPB provides analgesia to the anterolateral abdominal wall at the T6-L1 dermatomal levels and is commonly used for postoperative pain control after various abdominal surgeries, including laparoscopic cholecystectomy.

In this study, the investigators aim to compare the effectiveness of US-guided RIFPB and TAPB for postoperative pain management after laparoscopic cholecystectomy and to compare both techniques with a control group.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Scheduled for elective laparoscopic cholecystectomy

Exclusion Criteria:

* Known allergy to local anesthetics or opioid medications
* Infection at the planned block site
* History of alcohol or drug dependence
* Use of anticoagulant therapy
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | During the first 24 hours postoperatively
  Total postoperative opioid consumption will be recorded for each patient during the first 24 hours after surgery. Opioid use will be quantified based on the total dose of rescue opioid analgesics administered and compared between study groups to assess differences in postoperative opioid requirements.

SECONDARY OUTCOMES:
Postoperative pain scores | Postoperative hours 1, 3, 6, 12, 18, and 24.
  Postoperative pain will be assessed using the Numerical Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst pain imaginable. Pain scores will be recorded both at rest and during ambulation at 1, 3, 6, 12, 18, and 24 hours postoperatively. NRS scores will be compared between study groups to evaluate differences in postoperative pain intensity.
Adverse events | During the first 24 hours postoperatively
  Adverse events (nausea, vomiting, itching, ect) related to opioid use will be recorded for each patient
Postoperative Rescue Analgesic Consumption: | During the first 24 hours postoperatively
  The use of rescue analgesics in the postoperative period will be recorded and compared between study groups to evaluate differences in the need for additional analgesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Ciftci B, Omur B, Alver S, Akin AN, Yildiz Y, Tulgar S. The Medipol Combination: Novel Rectointercostal Fascial Plane Block and Pectointercostal Fascial Plane Block for Postoperative Analgesia Management After Cardiac Surgery: A Report of 15 Cases. A A Pract. 2024 Jun 5;18(6):e01794. doi: 10.1213/XAA.0000000000001794. eCollection 2024 Jun 1. PMID 38836555
- [Background] Dost B, Turunc E, Ozdemir E. Subxiphoid Pericardial Window Using a Combination of Rectointercostal Fascial Plane Block and Superficial Parasternal Intercostal Plane Block. J Cardiothorac Vasc Anesth. 2024 May;38(5):1282-1283. doi: 10.1053/j.jvca.2024.02.002. Epub 2024 Feb 4. No abstract available. PMID 38453556
- [Background] Tsai HC, Yoshida T, Chuang TY, Yang SF, Chang CC, Yao HY, Tai YT, Lin JA, Chen KY. Transversus Abdominis Plane Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:8284363. doi: 10.1155/2017/8284363. Epub 2017 Oct 31. PMID 29226150
- [Background] Brogi E, Kazan R, Cyr S, Giunta F, Hemmerling TM. Transversus abdominal plane block for postoperative analgesia: a systematic review and meta-analysis of randomized-controlled trials. Can J Anaesth. 2016 Oct;63(10):1184-1196. doi: 10.1007/s12630-016-0679-x. Epub 2016 Jun 15. PMID 27307177
- [Background] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789